CLINICAL TRIAL: NCT02475473
Title: Circulatory Levels of Irisin in Response to Chronic Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 504792B
Record Dates: First submitted 2015-02-03; First posted 2015-06-18 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The acute intervention will consist of 1 session of training following the program:
  Resistance Training Exercises. Each participant in the intervention group will perform resistance-training exercises in the form of a circuit. The circuit will consist of 10 repetitions per exercise of 7 exercises: leg press, bent-over row, bench press, squats, dumbbell jump squats with raises, dead-lifts and weighted abdominal crunches, with approximately 30 sec of rest in between each exercise (based on the estimated time needed to move from one position to the next). Initial intensity 6-7 of RPE and ending the set at 9-10. Each participant will move through the circuit 3 times, with 2 to 3 minutes of rest between each round.
  Interventions: Other: Exercise Training
- Control (No Intervention): Control

INTERVENTIONS:
Other: Exercise Training — Chronic High-Intensity Resistance Training
  Arms: Intervention

SUMMARY:
Study the responses of circulatory irisin to chronic high-intensity resistance training

DETAILED DESCRIPTION:
Objective: The purpose of this study is to study the circulating levels of irisin in response to chronic high-intensity resistance training in a group of healthy young adults.

Sample: The sample will be comprised 44 of adult men and women unpaid volunteers between the ages of 18 and 30.

Pre-screening assessments:

Informed consent, PAR-Q, Medical History and Exercise History will be used to determine health status and prior exercise experience. Menstrual cycle log will be required for female participants.

Pre-Intervention assessments:

* Anthropometric measurements and Body Composition: Height, triceps, thigh and calf skinfolds, biceps, thigh, hip, waist, and calf circumferences will be measured. Dual-energy x-ray absorptiometry (DEXA) will be performed to obtain body composition.
* Cardiopulmonary and Strength Fitness Testing. Cardiopulmonary fitness will be determined via maximum oxygen uptake testing. One maximum repetition (1-RM) will be used to assess the muscular fitness.
* Spontaneous Physical Activity: Daily activity level for 7 days will be collected.
* Familiarization. Participant will be instructed on the muscle conditioning techniques used for strength training so that the techniques can be mastered. The rate of perceived exertion (RPE) scale will also be used for familiarization during these sessions.

Intervention: The intervention will last 3 weeks with a frequency of 3 training session per week. We will collect blood samples levels at session 1 (at the beginning of week 1), session 3 (at the end of week 1), at session 6 (at the end of week 2) and session 9 (at the end of week 3). Blood draws will occur at the beginning of each session evaluated (pre-session), at the 45 min mark during each session and immediately after each session (post-session).

The sessions will consist on a circuit training of 3 sets of 7 exercises focused on major muscle groups. Ten repetitions on each circuit at 70% of the maximum capacity will be performed.

During the intervention:

- Blood-related variables. Baseline glucose, lactate and hematocrit will be obtained from all participants prior to intervention. Lactate and Hematocrit will be obtained pre-intervention and post-intervention, and within 1 min post workout at sessions 1, 3, 6 and 9.

Irisin will be obtained from blood samples at baseline, during and after training sessions 1, 3, 6 and 9. Irisin will be measured via a commercial enzyme-linked immunosorbent assay.

- Dietary Controls. Each participant will complete the Food Preference Questionnaire. In addition, the Automated Self-Administered 24-hour Recall (ASA24) will be collected for the days prior to sessions 1, 3, 6 and 9.

Post-Intervention assessments:

* Anthropometric measurements and Body Composition: Height, triceps, thigh and calf skinfolds, biceps, thigh, hip, waist, and calf circumferences will be measured. Dual-energy x-ray absorptiometry (DEXA) will be performed to obtain body composition.
* Caridorespiratory capacity determined via maximum oxygen uptake testing. One maximum repetition (1-RM) will be used to assess the muscular fitness.
* Spontaneous Physical Activity: Daily activity level for 7 days will be collected.

ELIGIBILITY:
Exclusion Criteria:

* Known health problems such as cardiovascular, pulmonary or metabolic disease will be excluded.
* Pregnant females.
* Any adults found taking medications that affect endocrine or cardiovascular function will also be excluded from the study.
* Individuals found to be less than 110 pounds.
* Participants that exercise more than three times per week or strength train more than twice per week.
* Individuals that have poor venous access or have expressed a fear of needles or having blood taken will also be excluded.
* Cigarette smoking (current or those who quit within the previous 6 months
* Hypertension
* Overweight and obese
* Pre-diabetics

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Serum irisin levels | Baseline and 3 weeks
Blood Lactate levels | 3 weeks
  Intensity of exercise on sessions 1, 3, 6 and 9
Changes in physical fitness levels as meassured by 1RM (repetition maximum) and Cardio-respiratory maximal testing | Baseline and 3 weeks
Changes in Body composition assessment: DEXA and anthropometry | Baseline and 3 weeks
Changes in Blood glucose levels | Baseline and 3 weeks
Changes in Hematocrit concentration | Baseline and 3 weeks
Diet assessment: 24 hour recall and Food Preference Questionnaire | 3 weeks
Physical Activity assessment: accelerometry | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez del Valle, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Exercise and Sport Sciences Building, Lubbock, Texas, United States